CLINICAL TRIAL: NCT07083193
Title: A Phase 1b, Multicenter, Open-label, Randomized Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of AC-101 Tablets in Participants With Moderate to Severe Active Ulcerative Colitis
Brief Title: A Study of AC-101 Tablets in Participants With Moderate to Severe Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Accro Bioscience (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC101-004
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AC-101 Dose 1 (Experimental): Participants will receive AC-101 Dose 1 as tablets orally twice daily from Week 0 through W12
  Interventions: Drug: AC-101
- AC-101 Dose 2 (Experimental): Participants will receive AC-101 Dose 2 as tablets orally once daily from Week 0 through W12
  Interventions: Drug: AC-101

INTERVENTIONS:
Drug: AC-101 — AC-101 tablets will be administered orally.

SUMMARY:
The purpose of the study is to evaluate the safety, efficacy, and pharmacokinetics of AC-101 tablets in participants with moderate-to-severe ulcerative colitis.

The total study duration is up to 17 weeks, including 4-week screening, 12-week treatment period, and 1-week safety follow-up.

The study will enroll approximately 24 participants with moderate to severe active ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ulcerative Colitis (UC) or suspected UC symptom for at least 3 months prior to enrolment and confirmed diagnosis of UC by endoscopic and histopathological examinations during screening.
* Evidence of active UC defined by modified Mayo score of 5 to 9 points (inclusive) with 3 subscores meeting the followings:

  1. Stool frequency (SF) subscore of .≥ 2 points, and
  2. Rectal bleeding (RB) subscore of .≥ 1 points, and
  3. Endoscopic (ES) subscore of ≥ 2 points (excluding friability), confirmed by screening endoscopy
* Disease extension of ≥ 15cm from anal verge, confirmed by screening endoscopy
* Currently using concomitant 5-salicylates (5-ASA) or oral corticosteroid (≤ 20 mg prednisone or equivalent, ≤ 9 mg budesonide MMX or equivalent) should keep stable doses from 2 weeks prior to enrolment till study completion.
* Biologic-naïve or previous biological treatment for more than 5 half-lives.

Exclusion Criteria:

* Previous/current documented diagnosis of Crohn's Disease (CD), indeterminate colitis, severe UC required hospitalization or corticosteroid pulse therapy, ulcerative proctitis, fulminant colitis, ischemic colitis and other intestinal diseases.
* Previous received 2 or more types of advanced treatment including biologics (e.g., TNF-α antibodies, IL-12/23 antibodies, integrin-α4β7 antibodies) and small molecule (e.g., JAK inhibitors, S1P receptor modulator), and all deemed by investigator as treatment failure.
* Intravenous/rectal administration of steroids or topical administration of 5-ASA within 2 weeks prior to enrolment; systemic administration of small molecule (e.g., Tofacitinib, Upadacitinib, Ozanimod) within 4 weeks prior to enrolment.
* Clostridium difficile infection or other enteric pathogen infection within 30 days prior to endoscopy, or positive for Clostridium difficile or other enteric pathogens prior to enrolment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events | Up to Week 13
  An Adverse Event (AE) is defined as any new untoward medical condition or worsening of a pre-existing medical condition following or during exposure to an investigation product, whether or not considered causally related to the product.

SECONDARY OUTCOMES:
Proportion of Participants Achieved Clinical Response | Week 12
  Clinical response is defined as achieving the following changes in the modified Mayo score (excludes the physicians' global assessment)
  1. A decrease from baseline in modified Mayo score of ≥ 2 points, and
  2. A decrease from baseline in modified Mayo score of ≥ 30%, and
  3. A decrease from baseline in rectal bleeding (RB) subscore of ≥ 1 point or absolute RB subscore ≤ 1 point
  The modified Mayo score is a sum of the following 3 subscores:
  1. Stool frequency (SF) subscore (0-3)
  2. Rectal bleeding (RB) subscore (0-3)
  3. Endoscopic (ES) subscore (0-3)
Proportion of Participants achieved Clinical Remission | Week 12
  Clinical remission is defined as achieving the following changes in the modified Mayo score
  1. Absolute modified Mayo score ≤ 2 points, and
  2. Absolute SF subscore ≤ 1 point, and
  3. Absolute RB subscore = 0 point, and
  4. Absolute ES subscore ≤ 1 point

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China